CLINICAL TRIAL: NCT02918305
Title: A Clinical Study of the Ultrasound Renal Denervation System in Patients With Resistant Hypertension
Brief Title: Renal Denervation on Quality of 24-hr BP Control by Ultrasound In Resistant Hypertension
Acronym: REQUIRE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: JIMRO Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RDN-15-001
Record Dates: First submitted 2016-09-27; First posted 2016-09-28 (Estimated); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Hypertension; Vascular Diseases
Keywords: denervation; resistant hypertension
MeSH Terms: conditions — Hypertension; Vascular Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- PRDS-001 Renal Denervation Ultrasound System (Sham Comparator): Randomization will occur following the diagnostic renal angiogram. Blinded patients randomized to treatment will receive the renal denervation procedure using PRDS-001 System to deliver ultrasound energy to thermally ablate and disrupt the renal sympathetic nerves while sparing the renal arterial wall.
  Interventions: Device: PRDS-001 Renal Denervation Ultrasound System
- Sham Procedure (Sham Comparator): Randomization will occur following the diagnostic renal angiography. For blinded patients randomized to control, the diagnostic renal angiography will be considered the sham procedure.
  Interventions: Procedure: Sham Procedure

INTERVENTIONS:
Device: PRDS-001 Renal Denervation Ultrasound System
  Other Names: renal denervation
  Arms: PRDS-001 Renal Denervation Ultrasound System
Procedure: Sham Procedure
  Other Names: renal angiography
  Arms: Sham Procedure

SUMMARY:
The REQUIRE STUDY is a multi-center, randomized, double-blind, sham-controlled study, which aims to confirm the efficacy and safety of PRDS-001 (ReCor Medical Inc. Paradise in Europe) for renal denervation therapy in patients with treatment resistance hypertension, in comparison with the sham procedure.

DETAILED DESCRIPTION:
Patients with treatment resistance hypertension is defined patients being treated on 3 or more different classes of antihypertensive medications including diuretics.

ELIGIBILITY:
Inclusion Criteria:

* average office systolic BP of 150 mmHg or greater or office diastolic BP of 90 mmHg or greater (both in the sitting position)
* 24-hr ambulatory BP 140 mmHg or greater.

Exclusion Criteria:

* Secondary hypertension (sleep apnoea can be included.)
* Type I diabetes or uncontrolled Type II diabetes with HbA1c 8.4% or greater
* Known or concurrent chronic active inflammatory bowel diseases (e.g. Crohn's disease, ulcerative colitis etc.)
* eGFR<40 mL/min/1.73m2 (per predictive equation Japanese Society of Nephrology)
* Known severe cardiovascular events within 3 months or severe cerebrovascular events
* Patients those who are planned to receive PCI or other operation for iscaemic cardiovascular disease within 8 months
* Concurrent persistent atrial fibrillation
* Patients those who are on active implantable medical devices
* Primary pulmonary hypertension
* Patients those who are contraindicated to, or confirmed to have intolerable anaphylactic reaction or uncontrollable allergy to contrast media

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2021-10 (Actual)

PRIMARY OUTCOMES:
a decrease of average 24-hr ambulatory systolic BP from the baseline | 3 month follow-up visit

SECONDARY OUTCOMES:
a decrease of the average ambulatory systolic BP during the daytime and that during the nighttime, from the baseline, respectively | 3 month follow-up visit
a decrease of the average ambulatory diastolic BP during the daytime, and that during the nighttime, from the baseline, respectively | 3 month follow-up visit
a decrease of the average office BP (both systolic and diastolic) in the sitting position from the baseline | 3 month follow-up visit

CONTACTS AND LOCATIONS:
Locations (53):
- Japan (44):
  - Hirosaki, Aomori
  - Urayasu, Chiba
  - Tōon, Ehime
  - Chikushino-shi, Fukuoka
  - Kasuga, Fukuoka
  - Kitakyushu, Fukuoka
  - Kurume, Fukuoka
  - Sekimachi, Gifu
  - Nayoro, Hokkaido
  - Sapporo, Hokkaido
  - Tomakomai, Hokkaido
  - Amagasaki, Hyōgo
  - Kobe, Hyōgo
  - Nishinomiya, Hyōgo
  - Kanazawa, Ishikawa-ken
  - Morioka, Iwate
  - Yokohama, Kanagawa
  - Kahoku, Kanazawa
  - Kōchi, Kochi
  - Suzuka, Mie-ken
  - Sendai, Miyagi
  - Nakagami, Okinawa
  - Kishiwada, Osaka
  - Sakai, Osaka
  - Suita, Osaka
  - Sayama, Saitama
  - Shimotsuke, Tochigi
  - Adachi City, Tokyo
  - Chiyoda City, Tokyo
  - Hachiōji, Tokyo
  - Meguro City, Tokyo
  - Minato, Tokyo
  - Minato-Ku, Tokyo
  - Musashino, Tokyo
  - Sakata, Yamagata
  - Fukuoka
  - Hiroshima
  - Kagoshima
  - Kumamoto
  - Kyoto
  - Miyazaki
  - Niigata
  - Okayama
  - Saga
- South Korea (9):
  - Busan
  - Daegu
  - Daejeon
  - Gangneung
  - Gwangju
  - Gyeonggi-do
  - Incheon
  - Seoul
  - Yangsan

REFERENCES:
- [Derived] Kario K, Yokoi Y, Okamura K, Fujihara M, Ogoyama Y, Yamamoto E, Urata H, Cho JM, Kim CJ, Choi SH, Shinohara K, Mukai Y, Ikemoto T, Nakamura M, Seki S, Matoba S, Shibata Y, Sugawara S, Yumoto K, Tamura K, Yoshihara F, Nakamura S, Kang WC, Shibasaki T, Dote K, Yokoi H, Matsuo A, Fujita H, Takahashi T, Kang HJ, Sakata Y, Horie K, Inoue N, Sasaki KI, Ueno T, Tomita H, Morino Y, Nojima Y, Kim CJ, Matsumoto T, Kai H, Nanto S. Catheter-based ultrasound renal denervation in patients with resistant hypertension: the randomized, controlled REQUIRE trial. Hypertens Res. 2022 Feb;45(2):221-231. doi: 10.1038/s41440-021-00754-7. Epub 2021 Oct 15. PMID 34654905